CLINICAL TRIAL: NCT04506359
Title: Develop and Test the Effects of the 'Computer-Assisted OPD Personalized Supportive Cancer Care Program (COPSCCP)' on Early Stage Lung Cancer Patients
Brief Title: Develop and Test the Effects of the 'Computer-Assisted OPD COPSCCP on Early Stage Lung Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 201401019RINC
Record Dates: First submitted 2018-12-03; First posted 2020-08-10 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Personalized Supportive Cancer Care Program; Physical symptom; Fear of cancer recurrence
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled clinical trial which to compare the short term and long-term effects of the COPSCCP vs. the control group as usual group on early stage lung cancer patients.
  For both groups, we assessed patients' outcomes (including baseline data) for 6 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, 12, 24 months after discharge from hospital).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple (Care Provider, Investigator, Outcomes Assessor) This study was not fully blinded; however, the group allocation was concealed from the patient and primary researcher until after baseline assessments were completed. A primary researcher obtained patient consent, collected selfreported assessments, and if the patients were randomized to intervention group, the intervention trainer explained the exercise program to participants. The study statistician and data managers remained blinded at all times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Control Group: Usual care +case manager care, UC group or Control group
- experimental group (Experimental): The experimental group is COPSCCP+ UC+ case manager care. In this group, a 6-month intervention providing for each time while subject visit their chest surgeon(s) in the OPD (from the first time before hospital discharge/T1) - usually patients visited hospital in 2 weeks, 1 month, 2 months, 3 months and 6 months (T2-6) after surgery. Patients will receive (a) nurse-guided touch-screen computer screening (assessment) for their psychological and physical distress and care needs during current week; (b) the screening /assessment results will immediately show as the outcome (we are developing a calculation system to sum those scores).
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Experimental Group — The Ex group is COPSCCP+ UC+ case manager care. In this group, a 6-month intervention providing for each time while subject visit their chest surgeon(s) in the OPD (from the first time before hospital discharge/T1).
  Arms: experimental group

SUMMARY:
Although there is a relatively better prognosis, the 5-year survival rate for early stage lung cancer (Stage I, II, IIIA) is still relatively low compared to those other types of cancer. These patients might suffer lots from the uncertainty and substantial disease and treatment related physical changes. The investigator aims to (1) Develop and construct the contents, related patient education materials and computerized systems of the three evidence and service-based lung cancer care programs, including (a) Control as usual care (UC+ case manager care, or Control group), and (b) Computer Assisted OPD Personalized Supportive Care Program (UC+COPSCCP or Ex group); and (2) Compare the effects of Ex and care as usual (receiving usual care and case manager care) on self-report quality of life (QOL), physical symptoms, physical function and fear of cancer recurrence (FCR) in newly diagnosed early-stage lung cancer patients. Eligible patients will be newly diagnosed early stage lung cancer patients (patients in stage I, II, & IIIA) who have received surgery. A 2-group randomized control trial (RCT) matching with cancer stages will be conducted. For the COPSCCP, patients will be intervened for 6 months from the first time during hospitalization of receiving surgery or before hospital discharge and then OPD intervention. Each patient will be followed 6 time points for 2 years (will be drop and refer to medical oncology while having recurrence, metastasis or death): baseline (pre-discharge from hospital) and 1, 3, 6, 12, and 24 months after discharge from hospital, T1-T6, respectively. The outcomes indicators will include: psychological variables, physical/disease variables, symptoms, lung function, and recurrence rate during 2 years. The estimated subjects would be 150 for each group, totally 300 subjects recruited in the beginning of the study. Results would be analyzed mainly by GEE and survival analysis. IRB approval will be received before the RCT. The investigator expects to develop and test the supportive cancer care interventions and generalize the interventions into the cancer care system after the study if prove good outcomes.

DETAILED DESCRIPTION:
Background: Although there is a relatively better prognosis, the 5-year survival rate for early stage lung cancer (Stage I, II, IIIA) is still relatively low compared to those other types of cancer. These patients might suffer lots from the uncertainty and substantial disease and treatment related physical changes. How to provide a feasible OPD personalized supportive care program is important.

Purpose: Main purpose of the study: (1) Develop and construct the contents, related patient education materials and computerized systems of the three evidence and service-based lung cancer care programs, including (a) Control as usual care (UC), and (b) Computer Assisted OPD Personalized Supportive Care Program (COPSCCP) (will be developed and structured the contents and computer system in the first 4 months of this research project); and (2) Compare the effects of COPSCCP and care as usual on self-report quality of life (QOL), physical symptoms, lung function, Depression, Anxiety, fear of recurrence, Unmet Cancer Needs, recurrence rate. Each patient will be follow for 2 years. Patients with recurrence, metastasis will be dropped out from the study (and refer to medical oncology).

Method: Eligible patients will be newly diagnosed early stage lung cancer patients (patients in stage I, II, & IIIA) who have received surgery. A 2-group randomized control trial (RCT) matching with cancer stages will be conducted. For the COPSCCP, patients will be intervened for 6 months from the first time during hospitalization of receiving surgery or before hospital discharge and then OPD intervention. Each patient will be followed 6 time points for 2 years (will be drop and refer to medical oncology while having recurrence, metastasis or death): baseline (pre-discharge from hospital) and 1, 3, 6, 12, and 24 months after discharge from hospital, T1-T6, respectively. The outcomes indicators will include: psychological variables, physical/disease variables, symptoms, lung function, and recurrence rate during 2 years. The estimated subjects would be 150 for each group, totally 300 subjects recruited in the beginning of the study. Results would be analyzed mainly by GEE and survival analysis. IRB approval will be received before the RCT. The investigator expects to develop and test the supportive cancer care interventions and generalize the interventions into the cancer care system after the study if prove good outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age ≥20 years
* early stage lung cancer
* had tumor excision surgery
* Mandarin / Chinese-reading and speaking

Exclusion Criteria:

* had double cancer
* had cancer recurrence or metastasis
* primary cancer unknown
* conscious unclear

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-04-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Quality of Life EORTC QLQ C30 | Outcome Assessments will be conducted for 6 times, the first time is at one day after tumor excision surgery (T1) and 2 weeks, 1 month, 2 months, 3 months and 6 months (T2-6) after surgery.
  Quality of life will be assessed by the EORTC-QLQ. This Instrument is consists of 30 items to measure three subscales, includes 2 items global health status/quality of life, 15 items functional domains and 13 items cancer common related symptoms or problems. Two items in global health status use a 7-point summated scale (1 = poor; 7 = excellent) and other items are rated on 4-point Likert's Scales (1=not at all; 4=very much). The scores will be transformed to a range from 0 to 100. In global health status and functional domains, the higher scores indicate better function. In the symptoms subscale, lower scores indicate less severe symptoms (Aaronson et al., 1993). The Taiwan Chinese version has been demonstrated to be both reliable and valid (Chie et al., 2004).
Changes in psychological distress | Outcome Assessments will be conducted for 6 times, the first time is at one day after tumor excision surgery (T1) and 2 weeks, 1 month, 2 months, 3 months and 6 months (T2-6) after surgery.
  The severity of lung cancer patients' anxiety and depression will be measured by the self-reporting HADS. The 14 items of HADS consists of two subscales, include 7 items anxiety and 7 items depression. The score of all items ranges from 0 (not at all) to 3 (always) and the total score of each subscale are ranged from 0 to 21, a higher score indicates a higher level of anxiety or depression. Satisfactory psychometrics of the HADS has been shown in cancer populations in Taiwan (Chen etal. 1999).
Changes in Fear of Recurrence | Outcome Assessments will be conducted for 6 times, the first time is at one day after tumor excision surgery (T1) and 2 weeks, 1 month, 2 months, 3 months and 6 months (T2-6) after surgery.
  The FoR-C is a Chinese version of the original FoR questionnaire1-3. The FoR questionnaire consists of six statements with a five-point response scale from not at all (1), a little, sometimes (2), a lot , and all the time) and one statement with a response scale from 0 (not at all) to 10 (a great deal). The summary of FoR was range from 6 to 40. Higher score indicates a higher level of fear of recurrence. The significance of the FoR was indicated by patients' responses 'a lot' or 'all the time' for the first six statements and the score of 7-10 for the last item, in which case. Current study will use the same approach to determine the cut-off point of the FoR.
Changes in Sleep Quality (SDQ) | Outcome Assessments will be conducted for 6 times, the first time is at one day after tumor excision surgery (T1) and 2 weeks, 1 month, 2 months, 3 months and 6 months (T2-6) after surgery.
  The quality of lung cancer patients' sleep will be measured by SDQ. The 12 items of SDQ was designed to evaluate patient' insomnia experience. Respondent score use a five-point Likert's scale (1 never true, 5 very often true) to indicate how often certain statements about insomnia. Higher scores reflect more dysfunctional beliefs about the causes and correlates of insomnia (Espie et al, 1989).
Changes in Brief Supportive Care Needs Survey (SCNS) | Outcome Assessments will be conducted for 6 times, the first time is at one day after tumor excision surgery (T1) and 2 weeks, 1 month, 2 months, 3 months and 6 months (T2-6) after surgery.
  The SCNS consists of 5 domains, include psychological, health system and information, daily living, patient care and sexuality domain. Response options "No need, not applicable (1); No need, satisfied (2); Low need (3); Moderate need (4); High need (5). The sum of item scores within each domain will be calculated and the scores will be transformed to a standardized score 0 to 100, higher score indicate moreunmet needs (Girgis et al, 2011). The higher scores representing more unmet needs. The Chinese SCNS34 has acceptable psychometric properties in previous lung cancer studies (Liao et al., 2011; Shun et al., 2014).
Changes in Muscle Power | Outcome Assessments will be conducted for 6 times, the first time is at one day after tumor excision surgery (T1) and 2 weeks, 1 month, 2 months, 3 months and 6 months (T2-6) after surgery.
  Patients' muscle strength (grip strength) of right and left hands will be assessed using Jamar Plus+ Digital Hand Dynamometer. Muscle endurance of right and left upper limbs and hip flexor muscle will be assessed using MicroFET2. Both grip strength meter and microFET 2 provided good reliability and validity for measuring muscle strength in the past studies. This measures has been applied in PI's currently head and neck study and early stage lung cancer follow up study.

CONTACTS AND LOCATIONS:
Overall Officials: Yeur-Hur Lai, Professor, Study Chair — School of Nursing, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Chie WC, Yang CH, Hsu C, Yang PC. Quality of life of lung cancer patients: validation of the Taiwan Chinese version of the EORTC QLQ-C30 and QLQ-LC13. Qual Life Res. 2004 Feb;13(1):257-62. doi: 10.1023/B:QURE.0000015295.74812.06. PMID 15058806
- [Background] Chen ML, Chang HK, Yeh CH. Anxiety and depression in Taiwanese cancer patients with and without pain. J Adv Nurs. 2000 Oct;32(4):944-51. PMID 11095234
- [Background] Espie CA, Brooks DN, Lindsay WR. An evaluation of tailored psychological treatment of insomnia. J Behav Ther Exp Psychiatry. 1989 Jun;20(2):143-53. doi: 10.1016/0005-7916(89)90047-5. PMID 2685045
- [Background] Girgis A, Lambert S, Lecathelinais C. The supportive care needs survey for partners and caregivers of cancer survivors: development and psychometric evaluation. Psychooncology. 2011 Apr;20(4):387-93. doi: 10.1002/pon.1740. Epub 2010 Apr 5. PMID 20878835
- [Background] Liao YC, Liao WY, Shun SC, Yu CJ, Yang PC, Lai YH. Symptoms, psychological distress, and supportive care needs in lung cancer patients. Support Care Cancer. 2011 Nov;19(11):1743-51. doi: 10.1007/s00520-010-1014-7. Epub 2010 Oct 15. PMID 20949362
- [Background] Shun SC, Yeh KH, Liang JT, Huang J, Chen SC, Lin BR, Lee PH, Lai YH. Unmet supportive care needs of patients with colorectal cancer: significant differences by type D personality. Oncol Nurs Forum. 2014 Jan 1;41(1):E3-11. doi: 10.1188/14.ONF.E3-E11. PMID 24368251